CLINICAL TRIAL: NCT01123863
Title: The Brigance Assessment Of Individual Neurodevelopment In Young Children With Sickle Cell Disease- 2
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRAIN2
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2015-06

CONDITIONS: Sickle Cell Disease
Keywords: Neuro cognitive deficits;; Brigance pre-school screen;
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient Group: This study will administer Brigance Preschool Screen -II to 3 year old children with SCD followed at St. Jude Children's Research Hospital
  Intervention: Brigance Preschool Screen -II
  Interventions: Other: Brigance Preschool Screen -II
- control group: The control group will consist of 3-year-old children attending day care in the Memphis area and serve as a population that come from a similar socioeconomic background as the SCD patient population.
  Intervention: Brigance Preschool Screen -II
  Interventions: Other: Brigance Preschool Screen -II

INTERVENTIONS:
Other: Brigance Preschool Screen -II — Three-year-old children with SCD who are followed at the St. Jude Children's Research Hospital Sickle Cell Center will be offered developmental screening with the Brigance Preschool Screen II during their regular clinic visits. Along with the screening test, socioeconomic data will be collected using a short questionnaire. Families will be asked to participate in this study by allowing us to collect their test results, medical information and socioeconomic data to compare with data collected from the control group. Parents who decline participation in this study will still be offered the Brigance Preschool Screen II as part of their child's clinical care.
  Groups: Patient Group
Other: Brigance Preschool Screen -II — Children in the Control Group will be given the Brigance preschool Screen-II Screening at the daycare they attend. The STARR coordinators have selected four daycare centers that have agreed to serve as control group sites. The family will be asked not to respond or aid the child during the assessment. One parent/guardian will fill out the Socioeconomic Data Collection Form while the examiner works with the child.
  The screening requires the child to give both verbal and non-verbal responses. The examiner records responses on the Three-Year-Old Child Data Sheet for the Brigance Preschool Screen-II. After the screening is complete the examiner collects the Socioeconomic Data Collection Form from the parent and leaves the room to score the assessment and write recommendations. The examiner then returns to the clinic room to discuss the results with the parent/guardian.
  Groups: control group

SUMMARY:
A preliminary study was conducted involving 88 three-year-old children with sickle cell disease (SCD) who were followed at the St. Jude Children's Research Hospital Sickle Cell Center. They were offered developmental screening with the Brigance Preschool Screen-II test during their regular clinic visits from January 2006 to August 2008. Data from this work showed that 50% of 3 year old children with SCD had low developmental screening scores. In addition, the low scores were found to be associated with less parental education and with speech deficits. However they were not associated with sickle cell genotype and hemoglobin level.

The primary goal of this study is to prospectively administer Brigance Preschool Screen -II to 3 year old children with SCD and 3 year old children without SCD who come from similar socioeconomic backgrounds and compare the results between the two groups.

DETAILED DESCRIPTION:
The primary objective of this study is to compare development in 3 year old children with SCD who are not on any treatment to age matched healthy controls using pass/fail rate for the Brigance Preschool Screen II.

Secondary objectives:

1. To compare the raw scores of the Brigance Preschool Screen II between SCD and control groups.
2. To compare the pass/fail rate and the raw scores between SCD patients who are not on any treatment and those who are being treated with hydroxyurea.
3. To compare the pass/fail rate and the raw scores between SCD patients on hydroxyurea treatment and the healthy controls
4. To assess the influence of medical factors on the Brigance Preschool Screen II performance in children with SCD.
5. To assess the influence of socioeconomic factors on the Brigance Preschool II results in children with SCD and controls.

ELIGIBILITY:
PATIENT GROUP

Inclusion criteria:

* 3.0-<4.0 years of age
* African-American
* Diagnosis of sickle cell disease (HbSS, HbSC, HbSβºthalassemia, HbSβ^+thalassemia)
* Followed at St. Jude Children's Research Hospital Sickle Cell Center

Exclusion criteria:

* Previous stroke
* Patients who are currently on a chronic transfusion program
* Known diagnosis associated with significant cognitive impairment (e.g. Down syndrome, mental retardation)
* Previously tested with Brigance Preschool Screen-II

CONTROL GROUP

Inclusion criteria:

* 3.0-<4.0 years of age
* African-American
* Attendee of day-care in Memphis area

Exclusion criteria:

1. Known diagnosis associated with significant cognitive impairment (e.g. stroke, Down syndrome, mental retardation)
2. Known diagnosis sickle cell disease (HbSS, HbSC, HbSβºthalassemia, HbSβ^+thalassemia)
3. Previously tested with Brigance Preschool Screen-II

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The patient group will consist of 3 year-old-children with SCD who are followed at the St. Jude Children's Research Hospital Sickle Cell Center. The control group will consist of 3-year-old children attending day care in Memphis.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2010-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Compare development in 3 year old children with SCD who are not on treatment to age matched controls using pass/fail rate for the Brigance Preschool Screen II. | 4 years

SECONDARY OUTCOMES:
Compare the raw scores of the Brigance Preschool Screen II between SCD and control groups. | 4 years
Compare the pass/fail rate and the raw scores between SCD patients who are not on any treatment and those who are being treated with hydroxyurea. | 4 years
Compare the pass/fail rate and the raw scores between SCD patients on hydroxyurea treatment and the healthy controls | 4 years
Assess the influence of medical factors on the Brigance Preschool Screen II performance in children with SCD. | 4 years
Assess the influence of socioeconomic factors on the Brigance Preschool II results in children with SCD and controls. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Estepp, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols